CLINICAL TRIAL: NCT01337349
Title: Effects of Pentoxiphylline on Left Ventricular Systolic Function Indices and Circulating Biomarkers in Patients With Chronic Congestive Heart Failure.
Brief Title: Effects of Pentoxiphylline on Left Ventricular (LV) Systolic Function Indices and Circulating Biomarkers in Patients With Chronic Congestive Heart Failure (CHF)
Acronym: PENT-CHF
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Did not enroll
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Karthikeyan Ananthasubramaniam, Director Nuclear Cardiology and Echocardiography, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2192010
Record Dates: First submitted 2011-04-15; First posted 2011-04-18 (Estimated); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Congestive Heart Failure
Keywords: Pentoxifylline; Chronic Congestive Heart Failure; Left Systolic Function; Biomarkers
MeSH Terms: conditions — Heart Failure | interventions — Pentoxifylline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sugar Pill (Placebo Comparator): Placebo control Group with sugar pill three times daily for 6 months
  Interventions: Drug: Placebo
- Pentoxifylline (Experimental): Pentoxifylline 400mg tablets to be taken three times daily for 6 months
  Interventions: Drug: Pentoxifylline

INTERVENTIONS:
Drug: Placebo — Sugar Pill 400mg taken orally three times a day for 6 months
  Arms: Sugar Pill
Drug: Pentoxifylline — Pentoxifylline 400mg taken orally Three times a day for 6 months
  Other Names: Trental
  Arms: Pentoxifylline

SUMMARY:
This is a prospective, double blinded randomized clinical study to evaluate the Effects of Pentoxifylline on left ventricular systolic function indices and circulating biomarkers in patients with chronic congestive heart failure.

A few studies all focused in Africa have consistently shown marked beneficial effects of pentoxifylline in improvement of left ventricular size and systolic function along with marked decrease in biomarkers of heart failure and apoptosis markers on top of standard CHF therapy. Furthermore pentoxifylline was shown to have negligible effects on heart rate, blood pressure in those studies. Limitations of these studies are that they are largely single center originating in the African subcontinent and have never been tested in the North American population, particularly Caucasians.

Despite major advances in medical therapy for congestive heart failure, it is still one of the leading causes of morbidity and mortality in North America. Most medications tested for improvement of Ejection Fraction with the exception of Beta-Blockers and Ace-Inhibitors have been associated with worsening mortality. Pentoxifylline is a medication that has negligible effects on myocardial oxygen consumption, yet promising effects on inflammatory markers seen in CHF with the possibility of improvement in LV systolic function and symptomology and may prove to be a useful addition for CHF patients. This would prove to be especially useful, particularly when associated with no major side effects.

DETAILED DESCRIPTION:
Patients who meet inclusion criteria will have a baseline physical exam, Heart Failure status assessment based on the Kansas City Heart Failure Questionnaire, EF assessment based on SPECT MUGA, cardiopulmonary exam to evaluate Vo2 max and assessment of left ventricular end diastolic and systolic dimensions based on 2D echo and labs drawn to assess circulating biomarkers. Patients will than be randomized into the control population where they will receive a placebo medication vs. the study population who will receive pentoxiphylline 400mg three times daily for 6 months. Patients will also have a one and three month clinic visit to assess for any potential change in symptoms and to assess medication compliance. Patients will then have a 6 month follow-up with repeat physical exam, Heart Failure status assessment based on the Kansas City Heart Failure Questionnaire, EF assessment based on SPECT MUGA, cardiopulmonary exam to assess Vo2 Max and assessment of left ventricular end diastolic and systolic dimensions based on 2D echo and labs drawn to assess circulating biomarkers.

ELIGIBILITY:
Inclusion Criteria:

1. Non-ischemic and ischemic class II-III heart failure patients on maximally tolerated evidence based medications. (i.e. BB (coreg, toprol, bisoprolol), ACEI/ARBS, Diuretics, +/- aldactone, digoxin).
2. Patients should also have an expected survival of greater than 6 months, including all other co-morbidities.
3. Sinus Rhythm
4. Age >18
5. LVEF <40% as assessed by (SPECT MUGA, ECHO).

Exclusion Criteria:

1. Class I and Class IV heart failure patients, patients who are newly diagnosed and currently are not on traditional evidence based medications.
2. Patients who have BiV-ICD placement.
3. Patients who decompensate into class IV heart failure during the study period requiring inotropes, LVAD, upgrade to BiV-ICD, will be reported on for potential treatment failure but will be taken out of the study.
4. Patients whose clinical conditions other than cardiomyopathy could influence inflammatory biomarkers. (i.e. Connective Tissue disorders, HIV)
5. Pregnancy
6. Severe exercise induced malignant ventricular arrhythmia
7. Any systemic process other than cardiomyopathy that would lead to survival <6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-07; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Improvement in Left Ventricular Ejection Fraction > 5% | 6 months
  Improvement in Left Ventricular Ejection Fraction > 5% (i.e: 20 to 25%) measured by SPECT MUGA after 6 months of pentoxifylline use.

SECONDARY OUTCOMES:
Left Ventricular End Systolic Volume Index | 6 months
  Improvement in Left Ventricular End Systolic Volume Index (decrease of 10%) as measured by 2D echo
Left Ventricular End Diastolic Volume Index | 6 Months
  Improvement in Left Ventricular End Diastolic Volume Index (decrease of 10%) as measured by 2D echo
Quality of Life Improvement | 6 Months
  Improvement in Quality of Life as Quantified by the Kansas City Heart Failure Questionaire.
Circulating Inflammatory Biomarkers | 6 Months
  Improvement in Circulating Inflammatory Biomarkers (e.g. TNF, IL6).
Change in VO2 Max | 6 Months
  Change in VO2 max over the study period. (With a change of 1 ml/kg/min as measured by cardiopulmonary exam considered meaningful.)

CONTACTS AND LOCATIONS:
Overall Officials: Karthikeyan Ananthasubramaniam, MD, Principal Investigator — Henry Ford Health Systems
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States